CLINICAL TRIAL: NCT02427360
Title: Evaluating the Efficacy of Artesunate-mefloquine on the Thai-Myanmar Border and the Relative Roles of Resistance Genetic Markers: A Retrospective Cohort Study
Brief Title: Evaluating the Efficacy of Artesunate-mefloquine and the Relative Roles of Resistance Genetic Markers
Acronym: MMA
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Texas Biomedical Research Institute (Unknown); Nanyang Technological University (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1409
Record Dates: First submitted 2015-04-22; First posted 2015-04-28 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: P. Falciparum Malaria; P. Falciparum Malaria Mixed Infection
Keywords: Retrospective Studies; Clinical Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective non randomized cohort to evaluate efficacy of MAS3 on patients with uncomplicated P. falciparum malaria or mixed infection (P. falciparum + a non-falciparum species). The review of patients' records and blood samples will be performed for patients treated at the clinics of Shoklo Malaria Research Unit from the period of January 2003 to December 2013.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the Day 42 PCR adjusted cure rate of mefloquine-artesunate (MAS3) in patients with P. falciparum

Study procedure

Clinic and patient records and log books will be reviewed and the following clinical information will be extracted: vital signs especially the temperature, clinical signs and symptoms, blood slide and haematocrit result and findings of physical examination (anaemia, jaundice, liver, spleen etc). As a routine, these data were recorded on the clinic patient record and malaria smear microscopy logbook accordingly (which will be regarded as the source documents in this analysis). These source documents will be reviewed and stored specimen will be analysed after getting the permission from the Director of Shoklo Malaria Research Unit, the University of Oxford Tropical Research Ethical Committee (OxTREC)and the Faculty of Tropical Medicine Ethics Committee (FTMEC). These data will be extracted and transcribed into the case record forms and entered into Microsoft access. During the data extraction, the unique ID will be assigned to each patient whereas the patients' name will neither be entered into database nor disclosed in the analysis process (ie: the data will be anonymised).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and sex who received treatment for uncomplicated malaria and followed up between January 2003 to December 2013
* Symptomatic of malaria infection, i.e. history of fever or tympanic temperature ≥37.5°c
* Microscopically confirmed asexual stages of P. falciparum ≥ 5/500 WBC (alone or mixed with non- P. falciparum species)
* Received fully supervised treatment of mefloquine-artesunate

Exclusion Criteria:

* Pregnant woman
* P. falciparum asexual stage parasitaemia greater than or equal to 4% red blood cells Signs or symptoms indicative of severe malaria29
* Mefloquine treatment within the 60 days preceding the current episode of malaria
* Splenectomy

Patients will be excluded from the efficacy analysis if they didn't finish the 3 days treatment of mefloquine artesunate but still kept in intention-to-treat population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with uncomplicated P.falciparum malaria or mixed infection (P.falciparum + a non-falciparum species) treated at the clinics of Shoklo Malaria Research Unit between 2003-2013. Medical records and stored/left-over samples from these patients will be reviewed/extracted and used for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
proportion of patients with clearance of asexual parasitaemia within 7 days of initiation of trial treatment | 42 days

SECONDARY OUTCOMES:
Proportion of aparasitaemic patients | day 3
gametocytaemia | 42 days
  gametocytaemia will be measured on pre and post treatment
haematocrit change | 42 days
  Haematocrit changes will be measured on pre and post treatment
Prevalence and temporal trend of resistance molecular markers | 42 days
  the following molecular markers will be measured; SNP on Kelch/K13 gene and Pfmdr1 copy number

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand